CLINICAL TRIAL: NCT07074392
Title: Assessing the Feasibility and Effect of Post-operative Electrical Stimulation on Spinal Accessory Nerve Recovery After Neck Dissection for Head and Neck Cancer
Brief Title: Assessing Spinal Accessory Nerve Recovery After Post-operative Electrical Stimulation
Acronym: SpARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19054
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Nerve Injury; Neck Dissection
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Electrical stimulation (Experimental): Post-operative electrical stimulation of spinal accessory nerve post neck dissection.
  Interventions: Device: Electrical Stimulation

INTERVENTIONS:
Device: Electrical Stimulation — Custom stimulator will deliver a 1hour stimulation protocol post-operatively at 20 Hz, with biphasic pulses (100 µs duration, 0-2mA amplitude range).
  Arms: Electrical stimulation

SUMMARY:
Shoulder weakness and pain are common after neck dissection surgery for head and neck cancer. This is often caused by injury to the spinal accessory nerve, which controls important shoulder muscles. Recovery can be slow and incomplete, affecting patients' ability to return to daily activities. This project will test whether a brief, low-dose electrical stimulation treatment can help the nerve heal faster and improve shoulder function. The treatment is applied during surgery and is safe, non-invasive, and quick to deliver. If successful, this approach could lead to better rehabilitation, less disability, and improved quality of life for patients undergoing cancer surgery. The project also supports the development of new medical technology and offers a pathway to expand the use of electrical stimulation in other nerve injuries.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing neck dissection

Exclusion Criteria:

* Previous neck dissection, previous implantable stimulator (i.e. pacemaker), previous spinal accessory nerve injury, pre-existing shoulder injury or weakness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Constant Murley Score (CMS) | 6 months post operative
  Shoulder function will be assessed using the Constant-Murley Score (CMS), a validated composite measure of shoulder function. The CMS ranges from 0 to 100 points, where higher scores indicate better shoulder function. The score incorporates four components: pain (15 points), activities of daily living (20 points), range of motion (40 points), and strength (25 points). A score of 100 represents full, pain-free shoulder function with normal strength and range of motion, while a score of 0 reflects complete dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Demographics Patient outcomes (CMS scores, electromyography and patient reported outcomes)

REFERENCES:
- [Result] Costello MC, Errante EL, Smartz T, Ray WZ, Levi AD, Burks SS. Clinical applications of electrical stimulation for peripheral nerve injury: a systematic review. Front Neurosci. 2023 Aug 3;17:1162851. doi: 10.3389/fnins.2023.1162851. eCollection 2023. PMID 37600003
- [Result] Gane EM, Michaleff ZA, Cottrell MA, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. Prevalence, incidence, and risk factors for shoulder and neck dysfunction after neck dissection: A systematic review. Eur J Surg Oncol. 2017 Jul;43(7):1199-1218. doi: 10.1016/j.ejso.2016.10.026. Epub 2016 Nov 17. PMID 27956321